CLINICAL TRIAL: NCT07294963
Title: Impact of Lifestyle Interventions on Cognitive Decline in NAFLD: A Randomized Controlled Trial of Liver Fibrosis, Hormonal Imbalance, and Inflammatory Markers
Brief Title: Impact of Lifestyle Interventions on Cognitive Decline in Non-alcoholic Fatty Liver Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: Northwest General Hospital and Research centre (Network); Khyber Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2025/010
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Neurocognitive Disorders
Keywords: Hepatocerebral Syndrome; Metabolic dysfunction-Associated SteatoHepatitis; Cognitive Decline; Liver Fibrosis; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Neurocognitive Disorders; Cognitive Dysfunction; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: A three-arm parallel-group randomized controlled trial will be conducted. Participants will be assigned to the Mediterranean Diet intervention, Control (general advice 2), and combined Mediterranean Diet + Structured Exercise intervention.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors conducting the Montreal Cognitive Assessment (MoCA) and laboratory technicians performing biomarker analyses (ELISA for T-Tau, cytokines, hormones) will be blinded to group assignment. Participants and the interventionists (dietitians, physiotherapists) cannot be blinded due to the behavioral nature of the lifestyle interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mediterranean Diet Intervention (Experimental): Participants will follow a structured, culturally adapted Mediterranean diet plan for 6 months, designed and supervised by a qualified dietitian. The diet emphasizes whole grains, vegetables, fruits, legumes, nuts, olive oil, and lean proteins (detailed 7-day plan in Annexure 7). Support includes individualized counseling, provision of meal plans, weekly food diaries, 24-hour dietary recalls, and monthly check-ins. Outcome assessments occur at T0, T1 (6 months), and T2 (12 months).
  Interventions: Behavioral: Structured Mediterranean Diet
- Control / General Advice (Active Comparator): Participants will receive general verbal and written advice on healthy eating and physical activity, consistent with standard care. No structured diet plan or supervised exercise will be provided. They will undergo all outcome assessments (FibroScan, FIB-4, MoCA, biomarker blood draws) at Baseline (T0), 6 months (T1), and 12 months (T2).
  Interventions: Behavioral: Control / General Advice
- Combined Diet and Exercise Intervention (Experimental): Participants will receive the identical Mediterranean diet intervention as Arm 2 plus a structured, progressive aerobic exercise program. The exercise consists of a 60-minute walking session, 5 days per week, for 6 months, progressing through conditioning, strength-building, and endurance phases (detailed in Annexure III). Compliance is monitored via exercise logs, fortnightly contact, and monthly check-ins. Outcome assessments occur at T0, T1 (6 months), and T2 (12 months).
  Interventions: Behavioral: Structured Mediterranean Diet; Behavioral: Control / General Advice

INTERVENTIONS:
Behavioral: Structured Mediterranean Diet — A culturally adapted, structured dietary plan based on the Mediterranean diet principles, delivered through individual dietitian counseling, provision of weekly meal plans, and ongoing compliance support (food diaries, recalls, monthly check-ins).
  Arms: Combined Diet and Exercise Intervention; Mediterranean Diet Intervention
Behavioral: Control / General Advice — This intervention consists of providing standardized, non-structured verbal and written information on the principles of a balanced diet and the benefits of regular physical activity, as per routine clinical practice. It serves as the active comparator representing minimal intervention.
  Arms: Combined Diet and Exercise Intervention; Control / General Advice

SUMMARY:
This study investigates whether a structured lifestyle program can help improve thinking skills and liver health in adults with Non-Alcoholic Fatty Liver Disease (NAFLD). We are enrolling 45 participants, aged 18-42, who will be randomly assigned to one of three groups for six months: one receiving general health advice, a second following a supervised Mediterranean diet plan, and a third combining the same diet with a regular walking program. The main goal is to see if these diet and exercise interventions can lead to better scores on memory and reasoning tests, reduce liver stiffness measured by a painless scan (FibroScan), and improve related blood markers of inflammation and hormone balance.

DETAILED DESCRIPTION:
This is a parallel-group, randomized controlled trial designed to evaluate the impact of lifestyle interventions on cognitive function in patients with NAFLD, and to explore associations with liver fibrosis severity and underlying biomarkers. The study aims to recruit 45 participants with imaging-confirmed NAFLD, who will be randomized (1:1:1) into a control group (general advice), a dietary intervention group (structured Mediterranean diet), or a combined intervention group (diet plus supervised exercise). Primary outcomes include cognitive performance measured by the Montreal Cognitive Assessment (MoCA) and serum T-Tau levels, assessed at baseline and after the 6-month intervention. Key secondary outcomes encompass changes in liver fibrosis (via FibroScan and FIB-4 index), inflammatory biomarkers (IL-6, TNF-α), and hormonal profiles (cortisol, testosterone, estradiol). The protocol has received ethical approval from the Khyber Medical University Institutional Review Board, and analysis will follow intention-to-treat principles using repeated-measures ANOVA and regression models to determine intervention efficacy and pathophysiological correlations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 42 years.
* Diagnosed with fatty liver (NAFLD) via imaging (e.g., ultrasound).
* Liver fibrosis assessed and staged via FibroScan and the FIB-4 index.
* Literate (to consent and complete cognitive assessments/questionnaires).

Exclusion Criteria:

* History of alcohol intake >20g/day.
* Chronic viral hepatitis B or C.
* Major neuropsychiatric illnesses.
* Pregnancy or breastfeeding.
* Chronic illnesses including Diabetes Mellitus and thyroid dysfunction.

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Composite of Heart Failure Hospitalization or Cardiovascular Death | From randomization up to study completion (maximum follow-up of 30 months).
  Time to first adjudicated event of either hospitalization for worsening heart failure or cardiovascular death. Events will be confirmed by a blinded Clinical Events Committee (CEC).
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score | Baseline, Month 12.
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item, self-administered disease-specific questionnaire. The Overall Summary Score (OSS) aggregates the physical limitation, symptom frequency, quality of life, and social limitation domains. Scores range from 0 to 100, where higher scores indicate better health status. The outcome is the change in KCCQ-OSS from baseline.
Change in N-terminal pro-brain natriuretic peptide (NT-proBNP) | Baseline, Month 6.
  The ratio of change in serum NT-proBNP level from baseline. NT-proBNP will be measured in pg/mL by a central laboratory using a standardized assay.
All-cause Mortality | From randomization up to study completion (maximum follow-up of 30 months).
  Time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ayesha Qaiser, PhD Scholar, Principal Investigator — Khyber Medical University Peshawar; Dr Inayat Shah, PhD, Principal Investigator — Institute of Basic Medical Sciences, Khyber Medical University; Dr Arshad Hussain, PhD, Principal Investigator — Northwest General Hospital, Peshawar
Locations (2):
- Pakistan (2):
  - Khyber Teaching Hospital, Peshawar, KPK
  - Northwest General Hospital, Peshawar, KPK

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in the primary publication (including demographic, clinical, laboratory, and cognitive assessment data) will be made available to qualified researchers upon reasonable request. The data will be shared to achieve the aims in the approved proposal, subject to a data use agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available 9 months after the publication of the primary results and will be accessible for 5 years.
Access Criteria: Data access requests should be directed to the corresponding author (Dr. Ayesha Qaiser) and will be reviewed by the trial's steering committee. Requestors will need to provide a methodologically sound proposal and sign a data use/access agreement.

REFERENCES:
- [Background] Kjaergaard K, Mikkelsen ACD, Wernberg CW, Gronkjaer LL, Eriksen PL, Damholdt MF, Mookerjee RP, Vilstrup H, Lauridsen MM, Thomsen KL. Cognitive Dysfunction in Non-Alcoholic Fatty Liver Disease-Current Knowledge, Mechanisms and Perspectives. J Clin Med. 2021 Feb 9;10(4):673. doi: 10.3390/jcm10040673. PMID 33572481
- [Background] Semmler G, Datz C, Reiberger T, Trauner M. Diet and exercise in NAFLD/NASH: Beyond the obvious. Liver Int. 2021 Oct;41(10):2249-2268. doi: 10.1111/liv.15024. Epub 2021 Aug 21. PMID 34328248
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Ishiba H, Sumida Y, Tanaka S, Yoneda M, Hyogo H, Ono M, Fujii H, Eguchi Y, Suzuki Y, Yoneda M, Takahashi H, Nakahara T, Seko Y, Mori K, Kanemasa K, Shimada K, Imai S, Imajo K, Kawaguchi T, Nakajima A, Chayama K, Saibara T, Shima T, Fujimoto K, Okanoue T, Itoh Y; Japan Study Group of Non-Alcoholic Fatty Liver Disease (JSG-NAFLD). The novel cutoff points for the FIB4 index categorized by age increase the diagnostic accuracy in NAFLD: a multi-center study. J Gastroenterol. 2018 Nov;53(11):1216-1224. doi: 10.1007/s00535-018-1474-y. Epub 2018 May 9. PMID 29744597